CLINICAL TRIAL: NCT05672550
Title: Dose-adjustment of Enoxaparin by a Bayesian Pharmacological Approach in Pediatric Kidney Transplant Recipients
Brief Title: Dose-adjustment of Enoxaparin by a Bayesian Pharmacological Approach in Pediatric Kidney Transplant Recipients (OPTI-TREX)
Acronym: OPTI-TREX
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180617; 2021-000099-12 (EudraCT Number)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Pediatric Kidney Transplant Recipients
Keywords: Kidney transplantation; Children; Enoxaparin; Bayesian based dose; Anti-Xa activity; allograft thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bayesian based dose adjustment (Experimental): Optimization of the enoxaparin dose using a bayesian program in order to prevent patients from complications due to the renal transplantation.
  A first recommended dose of enoxaparin (50 IU/kg) is administered subcutaneously during transplantation or within the first 24 hours.
  Then, in the experimental group, the dose is adjusted following a bayesian program integrated in the electronic Case Report Form which is based on each patient's data as the Anti-Xa activity
  Interventions: Drug: Bayesian based dose adjustment of enoxaparin
- Treatment as usual (empirical dose adjustment) (Active Comparator): Anti-Xa activity is measured and twice-daily enoxaparin empirical dose-adjustment is performed according to the usual practices in the investigating centers
  Interventions: Drug: Usual dose adjustment of enoxaparin

INTERVENTIONS:
Drug: Bayesian based dose adjustment of enoxaparin — A first recommended dose of enoxaparin 50 IU/kg subcutaneously is administered during transplantation or within the first 24 hours.
  Then a Bayesian estimate of individual pharmacokinetics is performed to adapt the next twice daily (Hour 12;Hour 24) enoxaparin dose until achievement of the target on two consecutive measurements. Then anti-Xa activity will be evaluated once a day until day 7.
  Arms: Bayesian based dose adjustment
Drug: Usual dose adjustment of enoxaparin — A first recommended dose of enoxaparin 50 IU/kg is administered during transplantation or within the first 24 hours. Then anti-Xa activity is measured and twice-daily (hour 12 ; hour 24) enoxaparin empirical dose-adjustment is performed according to the usual practices in the investigating centers to target.
  Arms: Treatment as usual (empirical dose adjustment)

SUMMARY:
Allograft vascular thrombosis is a devastating complication in kidney transplantation in adults and older children. Though uncommon, it is often irreversible and represents the main cause of graft loss within after kidney transplantation in adults and in the first post-operative year in children. Since allograft thrombosis is usually observed in the first 48h post-operatively, the need to promptly achieve appropriate anticoagulation in at-risk patients is of utmost importance.

However, no consensus exists regarding the optimal prophylaxis in the peri-transplant period and the following dose-adjustment, and practices are highly heterogeneous among centers. Moreover, the therapeutic target is very narrow and antithrombotic agents may conversely increase the risk of allograft hematoma. Enoxaparin is a low molecular weight heparin commonly used in this context, but off-label in children. Therapeutic ranges are based on anti-Xa levels 4 to 6 hours following injection and extrapolated from adults although evidences suggest that such extrapolation may be inappropriate in many circumstances. The current pediatric practice of dose adjustment to achieve and maintain a target anti-Xa range is empirical and dependent on the physician.

The aim of the proposed clinical trial is to assess the efficacy/safety profile of this bayesian-based dose optimization in the clinical setting, as compared to the current practices of empirical adjustment. This should greatly improve the personalized management of renal transplanted children, a subset of patients with singular renal function and little-investigated pharmacokinetics and help standardizing and rationalizing practices.

DETAILED DESCRIPTION:
The investigators will compare the efficacy of the Bayesian based dose versus the dose determined in a usual empirical way based on each physician's experience.

The primary endpoint is the Anti-Xa activity within the target range 28 to 30 hours after initiation of the treatment.

This is an open labelled randomized clinical trial. The randomization will proceed during the inclusion visit by the local pediatric nephrologist or intensivist just before the first enoxaparin injection, administered within 24 hours post-transplantation.

The investigators will conduct a national multicentric study with 9 inclusion centers which are all nephrology units specialized in renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric renal transplant recipients
2. Aged ≥ 2 years and ≤18 years
3. With an indication for enoxaparin treatment in the first post-transplant week according to the local transplant team such as inherited or acquired thrombotic disorders (eg. but not exclusive protein C, protein S, and antithrombin III deficiency; factor V Leiden mutation (FV506Q), prothrombin mutation (G20210A), mutation in the MTHFR (methyl Tetra hydro folate reductase) gene (C677T), and antiphospholipid antibodies (anticardiolipin antibodies and lupus anticoagulants), history of thrombosis, donor age < 2 years, recipient age < 5 years, cold ischemia time >24h, multiple renal vessels.
4. Informed consent form signed by the legal guardian(s)
5. Affiliated to a health insurance system, including AME

Exclusion Criteria

1. Per-transplant technical surgical problems
2. Pre-inclusion allograft thrombosis (before randomization and enoxaparin administration)
3. Peri-operative thrombosis or uncontrolled bleeding (before randomization and enoxaparin administration)
4. Peri-operative hemodynamic instability
5. Medical history of heparin-induced thrombocytopenia
6. Allergic reaction to enoxaparin or excipients
7. Pregnancy
8. LMWH (Low molecular weight heparins) prophylactic before transplant
9. UFH (unfractionated heparin) treatment during renal transplantation with an anti-Xa level detectable 4-6h post administration

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Anti-Xa activity within the target range | At 28-30 hours after initiation of treatment
  Anti-Xa activity within the target range (i.e., success defined by an anti-Xa activity ≥0.3 IU/mL and ≤0.5 IU/mL).

SECONDARY OUTCOMES:
Anti-Xa outcome measurement ≥0.3 IU/ml and ≤0.6 IU/mL | At 28-30 hours after initiation of treatment
  Anti-Xa outcome measurement is defined as: Anti-Xa activity 4-6 hours after the first enoxaparin injection on day 2
Difference between the Anti-Xa outcome measurement and the middle of the target range | At 28-30 hours after initiation of treatment
  Anti-Xa outcome measurement is defined as: Anti-Xa activity 4-6 hours after the first enoxaparin injection on day 2- the middle of the target range = 0.4UI/mL
Absolute difference between the Anti-Xa outcome measurement and the middle of the target range | At 28-30 hours after initiation of treatment
  Anti-Xa outcome measurement is defined as: Anti-Xa activity 4-6 hours after the first enoxaparin injection on day 2 - middle of the target range = 0.4UI/mL
Precision of Anti-Xa outcome measurement to reach the middle of the target range | At 28-30 hours after initiation of treatment
  Precision (Root Mean square Error) - middle of the target range = 0.4 UI/mL
Anti-Xa activity within the target range 4-6 hours after the 2nd enoxaparin injection | From 28-30 hours to 7 days after initiation of treatment
  Anti-Xa activity ≥0.3 IU/mL and ≤0.5 IU/mL
Anti-Xa activity ≥0.3 IU/mL and ≤0.6 IU/mL 4-6 hours after the 2nd enoxaparin injection | From 28-30 hours to 7 days after initiation of treatment
  Anti-Xa activity ≥0.3 IU/mL and ≤0.6 IU/mL
Time to achieve a target Anti-Xa activity (0.3-0.5 IU/mL) | From 28-30 hours to 7 days after initiation of treatment
  Time will be defined by the delay between date and time of treatment initiation and date and time of anti-Xa activity measurement in the target range.
Percentage of time within the target range | From 28-30 hours to 7 days after initiation of treatment
  The target range is defined as anti-Xa activity ≥0.3 IU/ml and ≤0.5 IU/mL from treatment initiation to D7 derived with individual predicted concentration time course
Graft thrombosis | Up to 30 days
  Graft thrombosis : assessed by allograft ultrasound
Enoxaparin-related side effects | Up to 30 days
  Enoxaparin-related side effects during the first postoperative month: bleeding (all localisations), graft hematoma (presence/absence): assessed by ultrasound
Allograft bleeding | Up to 30 days
  Allograft bleeding: bleeding with post-operative transfusion
Enoxaparin induced thrombopenia | Up to 30 days
  Thrombopenia

CONTACTS AND LOCATIONS:
Overall Officials: Olivia BOYER, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (10):
- France (10):
  - Hôpital Pellegrin, Bordeaux
  - CHU Félix Guyon, La Réunion
  - Hôpital Mère Enfant, Lyon
  - Hôpital de la Villeneuve, Montpellier
  - Hôtel Dieu, Nantes
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital des Enfants, Toulouse
  - Hôpital Necker - Enfants malades, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No